CLINICAL TRIAL: NCT04135482
Title: Evaluating the Immune Status of Patients With Severe Crohn's Disease Using Single Cell Sequencing
Brief Title: CD Patients Immune Status Evaluation
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: ZJU-JX-CD1
Record Dates: First submitted 2019-10-20; First posted 2019-10-22 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2019-10

CONDITIONS: Severe Crohn's Diease
Keywords: singcel cell sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Using the biospy samples of right colon or the last segment of ileum (both inflammation area and normal area nearby of 5cm), when patients receiving colonoscopy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CD: patients with severe crohn's disease
  Interventions: Other: colonic tissue biopsy

INTERVENTIONS:
Other: colonic tissue biopsy — colonic tissue biospy of patients with severe crohn's disease using colonoscopy

SUMMARY:
Using single cell sequencing method to evaluate and compare the immune status of patients with severe CD.

ELIGIBILITY:
Inclusion Criteria: 1, Patients with severe CD（CDAI>16,SES-CD>19） 2, Patients have no previous any drug therapy targeting CD or just received treatment of 5-ASA - Exclusion Criteria: 1, patients have previous treatment of prednisone, immunosuppressive agents such as azathioprine and biologic agents such as infliximab 2, patients were diagnozed as mild-moderate CD 3, patients have other immune disordered diseases such as SLE, PBC, AIH, PSC, sjogren syndrome, ulcerative colitis, and so on.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients were diagnosed as severe CD based on clinical, laboratory, endoscopic changes and imging.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
single cell analysis of the colonic tissue of patients with severe crohn's disease | 1 year
  single cell analysis of the colonic tissue of patients with severe crohn's disease: inflammed and non-inflammed area from right colon or the terminal ileum

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided